CLINICAL TRIAL: NCT02070913
Title: A Single-Center Case Series Clinical Study to Assess the Feasibility of Integrating Therapeutic Hypothermia Using the ZOLL IVTM System as an Adjunctive Therapy to Percutaneous Coronary Intervention in Patients With AMI
Brief Title: COOL-AMI EU Case Series Clinical Study
Status: Completed | Type: Observational
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Sponsor
Other Study IDs: EDC-2191
Record Dates: First submitted 2013-09-24; First posted 2014-02-25 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Hypothermia; Acute Myocardial Infarction; Percutaneous Coronary Intervention; AMI; PCI; Therapeutic Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A single-center, prospective case series clinical study consecutively enrolling up to 10 patients with expected duration of 12 months or less. The study objectives are to evaluate retention and the feasibility of integrating therapeutic hypothermia using the ZOLL IVTM System.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years of age.
* The patient must have symptoms consistent with AMI
* MI with ST-segment elevation
* The patient is eligible for PCI.
* The expected timing of the treatment pathway for the patient will allow for at least 10 minutes of cooling with the IVTM System prior to PCI.
* The patient or patient legal representative is willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

* The patient has had a previous myocardial infarction
* The patient is experiencing cardiogenic shock
* The patient is experiencing acute pulmonary edema.
* The patient is presenting with cardiac arrest.
* The patient is presenting with Killip risk stratification class II through IV.
* The patient is presenting with Atrial Fibrillation.
* The patient has a history of a prior large myocardial infarct or an infarct in the same segment that is currently affected.
* The patient requires an immediate surgical or procedural intervention other than PCI
* The patient has an aortic dissection.
* The patient has hepatic failure.
* The patient has end stage kidney disease.
* The patient is febrile
* Known chronic Congestive Heart Failure (CHF).
* Known previous CABG.
* Known recent stroke
* Cardio-pulmonary decompensation that has occurred en route to the hospital
* Contraindications to hypothermia
* The patient has a known hypersensitivity or contraindication to aspirin, heparin, or sensitivity to contrast media, which cannot be adequately pre-medicated.
* The patient has a known history of coagulopathy
* The patient is known to be pregnant
* The patient has a known hypersensitivity to antishivering medications.
* Patient has a known history of severe hepatic or renal impairment.
* The patient has an Inferior Vena Cava filter in place (IVC).
* The patient has a life expectancy of less than 1 year
* The patient has a known, unresolved history of drug use
* The patient is currently enrolled another investigational drug or device trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present with clinical signs and symptoms of acute myocardial infarction and meet all Inclusion and Exclusion criteria will be considered for case study presentation in this clinical trial without regard to age, gender or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2013-09; Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Time from hospital arrival to Percutaneous Coronary Intervention (PCI). | 24 hours
Time from hospital arrival to initiation of cooling. | 24 hours
Proportion of subjects achieving target temperature. | 24 hours

SECONDARY OUTCOMES:
Proportion of those enrolled that complete the study protocol. | 24 hours

CONTACTS AND LOCATIONS:
Locations (23):
- University Hospital Brno, Internal and Cardiology Department, Brno, Czechia
- North Estonia Medical Center, Tallinn, Estonia
- Ruppiner Kliniken GmbH, Neuruppin, Germany
- Hungary (8):
  - Heart Center Balatonfüred, Balatonfüred
  - Gottsegen Hungarian Institute of Cardiology, Budapest
  - Semmelweis University Heart and Vascular Center, Budapest
  - Medical Centre Hungarian Defence Forces, Budapest
  - Medical and Health Science Center University of Debrecen, Debrecen
  - University of Miskolc Borsod-Abauj-Zemplen County Hospital and University Teaching Hospital, Miskolc
  - Heart Institute University of Pecs, Pécs
  - Szent-Györgyi Albert Clinical Centre, II (University of Szeged), Szeged
- Vilnius University Hospital (Santariskiu Klinikos, Santariskiu), Vilnius, Lithuania
- Poland (4):
  - Nicolaus Copernicus University, Collegium Medicum University Hospital, Bydgoszcz
  - Medical University in Łódź, Bieganski Hospital, Lodz
  - Institute of Cardiology,, Warsaw
  - Silesian Center for Heart Diseases, Zabrze, Zabrze
- Serbia (3):
  - Clinical Center of Serbia Head of Department for invasive diagnostics (Division of Cardiology), Belgrade
  - Institute of Cardiovascular Diseases Vojvodina, Kamenitz
  - University Clinical Hospital Center Zemun, Zemun
- United Kingdom (4):
  - Royal Sussex County Hospital, Brighton
  - The London Barts Department of Cardiology, London
  - Cardiac Research Sister, King's College Hospital, London
  - Manchester Heart Centre Manchester Royal InfirmaryCentral Manchester University Hospitals NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided